CLINICAL TRIAL: NCT01318070
Title: A Phase 2/3, Double-Blind, Randomized, Placebo-Controlled, Parallel-Group, Multicenter Study to Determine the Efficacy and Safety of SYR-322 When Used in Combination With Thiazolidine in Subjects With Type 2 Diabetes in Japan
Brief Title: Efficacy and Safety of Alogliptin Used Combination With Thiazolidine in Participants With Type 2 Diabetes in Japan
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYR-322/CCT-004; UMIN000001382 (Registry Identifier: UMIN-CTR); JapicCTI-080590 (Registry Identifier: JapicCTI); U1111-1118-4073 (Registry Identifier: WHO)
Record Dates: First submitted 2011-03-16; First posted 2011-03-18 (Estimated); Results first posted 2011-07-06 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes Mellitus - Type2; Diabetes Mellitus; Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — alogliptin; Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Alogliptin 12.5 mg QD and Pioglitazone 15 or 30mg QD (Experimental)
  Interventions: Drug: Alogliptin and pioglitazone
- Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD (Experimental)
  Interventions: Drug: Alogliptin and pioglitazone
- Pioglitazone (15mg or 30mg ) QD (Active Comparator)
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Alogliptin and pioglitazone — Alogliptin 12.5mg, tablets, orally, once daily and Pioglitazone 15 or 30 mg, tablets orally once daily for up 12 weeks.
  Other Names: Alogliptin (SYR-322); Pioglitazone: Actos®
  Arms: Alogliptin 12.5 mg QD and Pioglitazone 15 or 30mg QD
Drug: Alogliptin and pioglitazone — Alogliptin 25 mg, tablets, orally, once daily and Pioglitazone 15 or 30 mg, tablets orally once daily for up 12 weeks.
  Other Names: Alogliptin (SYR-322); Pioglitazone: Actos®
  Arms: Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD
Drug: Pioglitazone — Pioglitazone 15 or 30 mg, tablets orally once daily for up 12 weeks.
  Other Names: Pioglitazone: Actos®
  Arms: Pioglitazone (15mg or 30mg ) QD

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of alogliptin, once daily (QD) combined with a thiazolidine taken QD in type 2 diabetic patients with uncontrolled blood glucose.

DETAILED DESCRIPTION:
Both insulin hyposecretion and insulin-resistance are considered to be involved in the development of type 2 diabetes mellitus.

Takeda is developing SYR-322 (alogliptin) for the improvement of glycemic control in patients with type 2 diabetes mellitus. Alogliptin is an inhibitor of the dipeptidyl peptidase IV (DPP-IV) enzyme. DPP-IV is thought to be primarily responsible for the degradation of 2 peptide hormones released in response to nutrient ingestion. It is expected that inhibition of DPP-IV will improve glycemic control in patients with type 2 diabetes.

The present study was planned to evaluate the efficacy and safety of alogliptin as an add-on to pioglitazone in type 2 diabetic patients with uncontrolled blood glucose despite treatment with pioglitazone as well as diet and exercise therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Had been taking pioglitazone at a stable dose (15 mg/day or 30 mg/day) for at least 16 weeks prior to the start of the treatment period (Week 0).
2. Had glycosylated hemoglobin (HbA1c) of 6.5% or more and below 10.0% at 14 weeks after the start of the observation period (Week -2).
3. Had HbA1c difference within 10.0%* at 10 weeks after the start of the observation period (Week -6) and 14 weeks after the start of the observation period (Week -2) from 10 weeks after the start of the observation period (Week -6) (*rounded off to the first decimal place).
4. Was receiving specific diet and exercise (if any) therapies during the observation period.

Exclusion Criteria:

1. Had taken a diabetic medications other than pioglitazone within 16 weeks before the start of the treatment period (Week 0).
2. Had a history or symptoms of cardiac failure.

Ages: 33 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 339 (Actual)
Dates: Start 2007-11; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Professor, Diabetes and Endocrine Division, Department of Medicine, Study Director — Kawasaki Medical School

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled at 33 investigative sites in Japan from 22 November 2007 to 22 October 2008.
Pre-assignment Details: Participants with historical diagnosis of type 2 diabetes with uncontrolled blood glucose despite treatment with pioglitazone as well as diet and exercise therapies were enrolled in one of 3, once-daily (QD) treatment groups.
Groups:
- Alogliptin 12.5 mg QD and Pioglitazone 15 or 30mg QD: Alogliptin 12.5mg, tablets, orally, once daily and Pioglitazone 15 or 30 mg, tablets orally once daily for up 12 weeks.
- Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD: Alogliptin 25 mg, tablets, orally, once daily and Pioglitazone 15 or 30 mg, tablets orally once daily for up 12 weeks.
- Pioglitazone 15 mg or 30 mg QD: Pioglitazone 15 or 30 mg, tablets orally once daily for up 12 weeks.
Period: Overall Study
Arm/Group | Alogliptin 12.5 mg QD and Pioglitazone 15 or 30mg QD | Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD | Pioglitazone 15 mg or 30 mg QD
Started | 111 | 113 | 115
Completed | 109 | 111 | 108
Not Completed | 2 | 2 | 7
Not completed — Adverse Event | 1 | 1 | 5
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Principal Investigator Discretion | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alogliptin 12.5 mg QD and Pioglitazone 15 or 30mg QD | Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD | Pioglitazone 15 mg or 30 mg QD | Total
Number analyzed (Participants) | 111 | 113 | 115 | 339
Age, Customized [Number; unit: participants]
  ≤ 64 years | 77 | 70 | 77 | 224
  ≥ 65 years | 34 | 43 | 38 | 115
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 43 | 39 | 126
  Male | 67 | 70 | 76 | 213

OUTCOME MEASURES:

1. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 2).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 2 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 2.
Population: Analysis based on last observation carried forward, where the last postbaseline double-blind observed value is carried forward and used for all subsequent scheduled time points where data is missing. Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD and Pioglitazone 15 or 30mg QD | Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD | Pioglitazone 15 mg or 30 mg QD
Number analyzed (Participants) | 110 | 111 | 115
percentage of Glycosylated Hemoglobin | -0.22 (0.150) | -0.22 (0.154) | -0.04 (0.186)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD and Pioglitazone 15 or 30mg QD vs Pioglitazone 15 mg or 30 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -0.179, 95% CI 2-sided [-0.224 to -0.135]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD vs Pioglitazone 15 mg or 30 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -0.180, 95% CI 2-sided [-0.225 to -0.135]

2. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 4).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 4 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 4.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD and Pioglitazone 15 or 30mg QD | Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD | Pioglitazone 15 mg or 30 mg QD
Number analyzed (Participants) | 111 | 113 | 115
percentage of Glycosylated Hemoglobin | -0.47 (0.236) | -0.46 (0.254) | -0.10 (0.301)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD and Pioglitazone 15 or 30mg QD vs Pioglitazone 15 mg or 30 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -0.363, 95% CI 2-sided [-0.434 to -0.292]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD vs Pioglitazone 15 mg or 30 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -0.359, 95% CI 2-sided [-0.432 to -0.287]

3. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 8).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 8 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 8.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD and Pioglitazone 15 or 30mg QD | Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD | Pioglitazone 15 mg or 30 mg QD
Number analyzed (Participants) | 111 | 113 | 115
percentage of Glycosylated Hemoglobin | -0.76 (0.353) | -0.81 (0.398) | -0.17 (0.433)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD and Pioglitazone 15 or 30mg QD vs Pioglitazone 15 mg or 30 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -0.588, 95% CI 2-sided [-0.692 to -0.484]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD vs Pioglitazone 15 mg or 30 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -0.635, 95% CI 2-sided [-0.743 to -0.526]

4. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 2).
Description: The change between the value of fasting plasma glucose collected at week 2 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 2.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Pioglitazone 15 or 30mg QD | Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD | Pioglitazone 15 mg or 30 mg QD
Number analyzed (Participants) | 110 | 113 | 115
mg/dL | -12.8 (14.68) | -17.0 (18.36) | -3.9 (18.25)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD and Pioglitazone 15 or 30mg QD vs Pioglitazone 15 mg or 30 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -8.83, 95% CI 2-sided [-13.20 to -4.47]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD vs Pioglitazone 15 mg or 30 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -13.06, 95% CI 2-sided [-17.86 to -8.26]

5. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 4).
Description: The change between the value of fasting plasma glucose collected at week 4 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 4.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Pioglitazone 15 or 30mg QD | Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD | Pioglitazone 15 mg or 30 mg QD
Number analyzed (Participants) | 111 | 113 | 115
mg/dL | -14.4 (18.45) | -17.9 (20.16) | -3.1 (19.54)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD and Pioglitazone 15 or 30mg QD vs Pioglitazone 15 mg or 30 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -11.24, 95% CI 2-sided [-16.22 to -6.25]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD vs Pioglitazone 15 mg or 30 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -14.82, 95% CI 2-sided [-20.00 to -9.63]

6. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 8).
Description: The change between the value of fasting plasma glucose collected at week 8 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 8.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Pioglitazone 15 or 30mg QD | Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD | Pioglitazone 15 mg or 30 mg QD
Number analyzed (Participants) | 111 | 113 | 115
mg/dL | -17.1 (16.96) | -21.3 (20.20) | -4.2 (22.29)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD and Pioglitazone 15 or 30mg QD vs Pioglitazone 15 mg or 30 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -12.88, 95% CI 2-sided [-18.09 to -7.68]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD vs Pioglitazone 15 mg or 30 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -17.08, 95% CI 2-sided [-22.64 to -11.53]

7. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 12).
Description: The change between the value of fasting plasma glucose collected at week 12 or final visit and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 12.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Pioglitazone 15 or 30mg QD | Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD | Pioglitazone 15 mg or 30 mg QD
Number analyzed (Participants) | 111 | 113 | 115
mg/dL | -14.9 (18.42) | -18.9 (20.96) | -2.4 (26.84)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD and Pioglitazone 15 or 30mg QD vs Pioglitazone 15 mg or 30 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -12.46, 95% CI 2-sided [-18.51 to -6.40]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD vs Pioglitazone 15 mg or 30 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -16.49, 95% CI 2-sided [-22.78 to -10.19]

8. Secondary Outcome: Change From Baseline in Blood Glucose Measured by the Meal Tolerance Test (Week 12).
Description: The change between the value of blood glucose measured by the meal tolerance test collected at week 12 or final visit and blood glucose measured by the meal tolerance test collected at baseline. Meal tolerance test measures blood glucose through blood samples drawn before a meal and 2 hours after the start of the meal.
Time Frame: Baseline and Week 12.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Pioglitazone 15 or 30mg QD | Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD | Pioglitazone 15 mg or 30 mg QD
Number analyzed (Participants) | 110 | 111 | 109
mg/dL | 58.3 (28.75) | 49.4 (29.27) | 70.6 (39.58)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD and Pioglitazone 15 or 30mg QD vs Pioglitazone 15 mg or 30 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -12.31, 95% CI 2-sided [-21.51 to -3.10]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD vs Pioglitazone 15 mg or 30 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -21.19, 95% CI 2-sided [-30.43 to -11.95]

9. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 12).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 12 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 12.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD and Pioglitazone 15 or 30mg QD | Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD | Pioglitazone 15 mg or 30 mg QD
Number analyzed (Participants) | 111 | 113 | 115
percentage of Glycosylated Hemoglobin | -0.91 (0.441) | -0.97 (0.517) | -0.19 (0.552)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD and Pioglitazone 15 or 30mg QD vs Pioglitazone 15 mg or 30 mg QD; Test type: Superiority or Other; Median Difference (Final Values) = -0.717, 95% CI 2-sided [-0.848 to -0.586]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD vs Pioglitazone 15 mg or 30 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -0.773, 95% CI 2-sided [-0.913 to -0.634]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are any unfavorable and unintended sign, symptom or disease temporally associated with the use of a medicinal product reported from first dose of study drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Alogliptin 12.5 mg QD and Pioglitazone 15 or 30mg QD | Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD | Pioglitazone 15 mg or 30 mg QD
Serious Adverse Events (participants affected / at risk) | 1/111 | 2/113 | 5/115
Other Adverse Events (participants affected / at risk) | 5/111 | 17/113 | 13/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alogliptin 12.5 mg QD and Pioglitazone 15 or 30mg QD (N=111) | Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD (N=113) | Pioglitazone 15 mg or 30 mg QD (N=115)
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alogliptin 12.5 mg QD and Pioglitazone 15 or 30mg QD (N=111) | Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD (N=113) | Pioglitazone 15 mg or 30 mg QD (N=115)
Nasopharyngitis (Infections and infestations) | 5 | 13 | 6
Dental caries (Gastrointestinal disorders) | 0 | 0 | 4
Blood creatine phosphokinase increased (Investigations) | 0 | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The clinical trial contract states that information should never be disclosed without prior consent of the sponsor, although it does not specify the number of days during which disclosure of information is limited.